CLINICAL TRIAL: NCT04351048
Title: The Evaluation of Stepwise and One Step Excavation Techniques In The Management of Deep Dentin Lesions
Brief Title: Stepwise and One Step Techniques In Deep Dentin Lesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: TIJEN PAMIR (Other)
Responsible Party: Sponsor-Investigator, TIJEN PAMIR, Prof Dr, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 70198063-050.06.0416-12.1/12
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Dental Caries, Dental Pulp Exposure
Keywords: Selective Caries Removal; Deep Dentin Lesion; Permanent Teeth; Stepwise and One Step Excavation Technique
MeSH Terms: conditions — Dental Caries; Dental Pulp Exposure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SW (Experimental): stepwise excavation
  Interventions: Procedure: Stepwise Excavation
- OneS (Experimental): one step excavation
  Interventions: Procedure: One Step Excavation

INTERVENTIONS:
Procedure: Stepwise Excavation — * stepwise excavation includes selective caries removal to soft dentine on pulpal wall in the first stage of the excavation and
  * after six months, the second stage of intervention includes re-entring the cavities and wall selective removal to firm dentine on pulpal wall.
  Arms: SW
Procedure: One Step Excavation — *one step excavations is completed in the first stage via performing selective removal to soft dentine on pulpal wall of the cavities.
  Arms: OneS

SUMMARY:
This double blind, randomized, controlled clinical trial aimed to observe the success of stepwise (SW) and one step (OneS) excavation techniques in the management of deep dentin caries. Additionally, evaluation of glass ionomer cement (GIC) as temporary restorative was also performed. For this purpose, forty participants were selected among the routine patients coming to university clinic. A permanent tooth having caries lesions penetrating to 75 percentage or more of dentin of patient were included. Randomization to SW and OneS groups were organized by coin method. The periphery of the cavities including enamel-dentin junction was cleaned until reach to hard dentin. Afterwards, selective removal to soft dentin on the pulpal side of the cavities was applied manually excavation and covered with pure calcium hydroxide and zinc oxide eugenol cement. GIC was used for temporary filling. This process was implemented both the first stage excavation of SW and OneS groups. Clinical and radiographic evaluations were performed at 6 months according to clinical signs and symptoms and radiographic sings using Periapical Index (PAI). Besides, temporary restorations were evaluated according to the of Ryge/Modified USPHS criteria. Following this evaluation, on the SW group, the cavities was re-entered and selective removal was applied up to firm dentin and pulp-capping were applied as mentioned above. In OneS group, temporary restoration was reduced as a base. All of the cavities were permanently restored with resin composite. Whole procedure was completed at one centre by a specialist, and control sessions was performed two experienced experts. Participants and experts were blinded in this study.

ELIGIBILITY:
Inclusion Criteria:

* Molar teeth with primary caries lesion prolonged of 75 percentage or more of dentin radiographically1 Existence of vitality with positive response to

  * electrical pulp test and
  * cold test
* No history of spontaneous pain on the teeth
* No sign of pain on percussion and palpation (sensitivity)

Exclusion Criteria:

* Individuals with the systemic disease who require hospitalization (oncological treatment, transplantation patients)
* Patients with uncontrolled hyperglycaemia or using insulin
* Patients with pregnancy/suspected
* Observation of radiolucency in the apex of the relevant tooth (PAI> 2)
* Secondary decayed teeth

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Pulpal Success Assessment | a 6-month periods
  Presence of vitality in treated tooth with positive response to electrical and thermal stimuli, no history of spontaneous pain and no response to percussion and pain (sensitivity) sign in palpation
Health Status of Periapical Tissue | a 6-month periods
  According to Orstavik' Periapical Index (PAI),
  Periapical Index score scale are 1to 5 :
  scoring with PAI 1 or PAI 2 refer to healthy tooth but PAI 3, PAI 4 and PAI 5 as worse outcome for periapical tissue that sing of periapical tissue damage

CONTACTS AND LOCATIONS:
Overall Officials: Tijen Pamir, Ph.D, Study Director — Ege University

REFERENCES:
- [Background] Innes NP, Frencken JE, Bjorndal L, Maltz M, Manton DJ, Ricketts D, Van Landuyt K, Banerjee A, Campus G, Domejean S, Fontana M, Leal S, Lo E, Machiulskiene V, Schulte A, Splieth C, Zandona A, Schwendicke F. Managing Carious Lesions: Consensus Recommendations on Terminology. Adv Dent Res. 2016 May;28(2):49-57. doi: 10.1177/0022034516639276. PMID 27099357
- [Background] Bjorndal L, Reit C, Bruun G, Markvart M, Kjaeldgaard M, Nasman P, Thordrup M, Dige I, Nyvad B, Fransson H, Lager A, Ericson D, Petersson K, Olsson J, Santimano EM, Wennstrom A, Winkel P, Gluud C. Treatment of deep caries lesions in adults: randomized clinical trials comparing stepwise vs. direct complete excavation, and direct pulp capping vs. partial pulpotomy. Eur J Oral Sci. 2010 Jun;118(3):290-7. doi: 10.1111/j.1600-0722.2010.00731.x. PMID 20572864
- [Background] Maltz M, Jardim JJ, Mestrinho HD, Yamaguti PM, Podesta K, Moura MS, de Paula LM. Partial removal of carious dentine: a multicenter randomized controlled trial and 18-month follow-up results. Caries Res. 2013;47(2):103-9. doi: 10.1159/000344013. Epub 2012 Nov 28. PMID 23207420
- [Background] Hayashi M, Fujitani M, Yamaki C, Momoi Y. Ways of enhancing pulp preservation by stepwise excavation--a systematic review. J Dent. 2011 Feb;39(2):95-107. doi: 10.1016/j.jdent.2010.10.012. Epub 2010 Dec 3. PMID 20971154